CLINICAL TRIAL: NCT06558305
Title: Effect of cDMARD and Baricitinib Therapy on IL-6, IL-12, IL-15 and IL-23 Expression Levels in Rheumatoid Arthritis Patients
Brief Title: IL-6, IL-12, IL-15 and IL-23 Expression Levels in Rheumatoid Arthritis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Sayed Ibrahim Abdelrahman, principal investigator, Assiut University
Other Study IDs: Interleukins in RA patients
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients on cDMARDS
  Interventions: Other: blood sample
- Patients on janus kinase (JAK) inhibitors
  Interventions: Other: blood sample
- Control
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — Total RNA will be extracted from the whole blood using a commercial extraction kit (RNA Extraction Kit, applied biotechnology Co.Ltd, Egypt) according to the manufacturer's instructions. RNA will be stored at -80°C.The extracted RNA will be used for cDNA synthesis using commercial kits (cDNA Synthesis Kit, applied biotechnology Co.Ltd, Egypt), according to the manufacturer's instruction.

SUMMARY:
Rheumatoid Arthritis (RA) is a systemic autoimmune disease characterized by chronic inflammation and articular damage.

Continuous medical research has dramatically improved the outcomes for patients with RA. Traditional therapeutic approaches have relied on glucocorticoids, nonsteroidal anti-inflammatory drugs (NSAIDs) and disease modifying antirheumatic drugs (DMARDs) such as methotrexate, sulfasalazine or leflunomide. Glucocorticoids and NSAIDs interfere with the inflammatory cascades while DMARDs impede both the inflammatory and the destructive processes of RA.

These drugs, although efficient, are not specifically directed against inflammatory cells or cytokines and are associated with significant toxicity. The development of biologic DMARDs (bDMARDs), has been an important step forward. Their ability to neutralize specific cytokines or target distinct immune cells filled a gap in existing treatment options for RA. [3]. However, some patients still have only partial or no response to bDMARDs. More recently, a group of drugs has been developed that inhibit the janus kinase (JAK) family of intracellular tyrosine kinases, which transmit cytokine- mediated signals via the JAK-signal transducer and activator of transcription (STAT) pathway [4]. Baricitinib, with a selectivity to inhibit JAK1 and 2, has been FDA approved for RA in 2018 [5].

Many cytokines such IL-6, IL-12, IL-15, IL-23, (GM-CSF) and (IFNs) are associated with the pathogenesis of RA. These cytokines transduce signals via the JAK-STAT pathway.

ELIGIBILITY:
Inclusion Criteria:

* Age is at leasr18 years old,
* established RA diagnosis according to 2010 the American College of Rheumatology/European League against Rheumatism classification criteria

Exclusion Criteria:

* Associated autoimmune diseases,
* connective tissue diseases,
* chronic liver or kidney diseases or
* genetic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: this study will include 30 RA patients receiving cDMARDs, 30 RA patients receiving baricitinib and 20 healthy participants.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
assess the effect of cDMARD and Baricitinib (JAKi) therapy on gene expressions of IL-6, IL-12, IL-15 and, IL-23 in patients with RA relative to the healthy controls. | 6 months
  assess the effect of cDMARD and Baricitinib (JAKi) therapy on gene expressions of IL-6, IL-12, IL-15 and, IL-23 in patients with RA relative to the healthy controls.

IPD SHARING:
Plan to Share IPD: Undecided